CLINICAL TRIAL: NCT05636020
Title: Intervention to Change Affect Recognition and Empathy (ICARE)
Brief Title: Intervention to Change Affect Recognition and Empathy
Acronym: ICARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Flora Hammond, Department Chair of Physical Medicine and Rehabilitation, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16937
Record Dates: First submitted 2022-11-22; First posted 2022-12-05 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Traumatic Brain Injury; Concussion, Intermediate; Concussion, Severe; Concussion With LOC 31 to 59 Minutes; Concussion With Brief Loss of Consciousness; Traumatic Brain Injury With Brief Loss of Consciousness; Traumatic Brain Injury With Loss of Consciousness; Traumatic Brain Injury With Prolonged Loss of Consciousness; Traumatic Brain Injury (TBI); Concussion, Initial Encounter; Traumatic Brain Injury (TBI); Concussion, Subsequent Encounter; Traumatic Brain Injury With No Loss of Consciousness; Traumatic Brain Injury With Open Intracranial Wound; Traumatic Brain Injury With Moderate Loss of Consciousness
Keywords: brain injury; affect recognition; empathy; caregiver; interpersonal behaviors; relationship closeness; mood; teletherapy; social cognition; theory of mind; perspective taking
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (ICARE) (Experimental): ICARE treatment consisting of 12 sessions that train affect recognition and empathic behaviors.
  Interventions: Behavioral: ICARE Treatment

INTERVENTIONS:
Behavioral: ICARE Treatment — The treatment is 12 teletherapy sessions lasting approximately 60-90 minutes. Of the 12 treatment sessions, 7 of them will focus on training skills to help the participant with TBI better recognize emotions from facial expressions. The remaining 5 sessions will teach skills important for empathizing with others' thoughts and feelings, and how to be emotionally supportive. Role-playing will be a big part of these last 5 sessions. The care-partner will be expected to attend as many of these 5 empathy sessions with the participant with TBI as possible.

SUMMARY:
Determine the feasibility, practicality, and early efficacy of a TeleRehab program (ICARE) to improve outcomes for persons with traumatic brain injury (TBI) in recognizing and responding to others' emotions alongside their care partner (CP).

DETAILED DESCRIPTION:
This phase I proof of principle pilot study of ICARE will be a non-randomized, one-group pre/posttest design with a double pretest, and an immediate posttest, with 3 and 6-month follow-ups in 40 participants with TBI and their CP. The study objectives are to explore the feasibility, practicality and early efficacy of ICARE to improve affect recognition (AR), empathy, interpersonal behaviors, and participation for persons with TBI. For CPs, goals are for them to feel more emotionally supported by the person with TBI; feel more in control of their own emotions, and have less CP anxiety. An additional objective for both participants with TBI and the CP is to enhance the quality and closeness of their relationship. For both TBI and CP participants, we anticipate ICARE will have good feasibility and acceptability, and post-treatment assessments will show significant improvements in perceived relationship closeness and relationship quality. For the TBI participants, we anticipate the post-treatment assessments will show significant improvements in affect recognition, empathy, interpersonal behavior, participation, and global impression of change. For the CPs, we anticipate the post-treatment assessments will show significant improvements in perceived emotional support (received from participant with TBI); suppression of self-emotions; and self-rated anxiety.

ELIGIBILITY:
Inclusion Criteria for TBI participant:

* Mild, moderate, or severe TBI determined by The Ohio State University Traumatic Brain Injury Identification Method (OSU TBI-ID) during Time 1; if mild, must have been at least dazed and confused. Must be ≥ 1-year post-TBI (unlikely spontaneous recovery). Must have a care-partner (CP) willing to participate. Must either have a ≤ 45 T score on any one of the SASNOS Interpersonal Behavior subscales or Total Interpersonal behavior score, OR select never, rarely, or occasionally to #2, #6, #7, and/ or #12 (obtained during screening process). Also, either: A) Must be believed by person with TBI OR B) Person with TBI has been told by others OR CP, that their problems with recognizing and/ or empathizing with others' emotions (self or CP rated) are believed to be new or worse since TBI and impacting their interpersonal behaviors or relationships.

Inclusion Criteria for CP:

* Must be a relative, spouse, or friend who believes the have sufficient interactions (~3 times/ week) with the participant with TBI to judge their empathic, interpersonal, and other behaviors. Must be willing to participate in assessments and empathy sessions.

Inclusion Criteria for both TBI and CP:

* Must be ≥18 years old. Must be a U.S. resident (exclusion for California residents). Must be proficient in English; have basic comprehension & ability to follow directions (determined via interaction at screening); have access to a computer or tablet with reliable internet (capacity for video conferencing) with video-conferencing capability.

Exclusion Criteria for TBI participant:

* Any other formal neurological disorder or condition that impacts emotional functioning other than TBI (e.g., stroke); suicide risk determined to be >low risk based on PI discretion and/or results of suicide protocol (if triggered); unstable or anticipated medication changes that will influence mood/ affect during study participation; and individuals who recently started psychotherapy (e.g., < 3 months ago) and/or active treatment in family or couples therapy.

Exclusion Criteria for CP:

* Moderate to severe TBI determined by the "OSU TBI-ID + ABI" (i.e., scoring a 4 or 5 on Worst Injury Scale); If the person indicates a mild TBI (OSU score of 2 or 3) or any other neurological impairment on the OSU (e.g. a stroke), then the person will be asked follow-up questions to determine if there were any persistent changes in thinking, memory, mood, social functioning that they believe was a result of the injury. PI and/ or Co-PI discretion will be used to evaluate the answer and determine inclusion or exclusion.

Exclusion Criteria for both TBI and CP:

* Developmental; neurodegenerative; major psychiatric disorder (e.g., schizophrenia, personality disorder); visual, hearing, or communication deficits that would impede participation; participation in IRB#12561; contemplating separation or divorce with the dyad partner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in St. Andrew's Swansea Neurobehavioral Outcome Scale-Interpersonal Behavior (SASNOS-IB) | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  Behaviors and symptoms of neurobehavioral dysfunction are rated on items covering 5 major domains, one of which is interpersonal behavior, which has 3 subdomains (social interactions, relationships, engagement). Prevalence of behaviors are rated using a 7-point scale ('never' to 'always'). Participants with TBI and CP will only complete the Interpersonal Behavior (IB) domain about the person with TBI. Psychometric property testing indicated excellent discriminant validity and good test-retest reliability.

SECONDARY OUTCOMES:
Change in The Diagnostic Assessment of Nonverbal Accuracy-2, Adult Faces (DANVA2-AF) | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (TBI participant only) The DANVA2-AF is a standardized performance-based measure of facial affect recognition. Participants will be shown 24 photographs of 4 facial expressions (different faces from ICARE training) and required to select a response option from a list of choices. Scores range from 0-24. The DANVA2-AF has high internal consistency, test-retest reliability, and good convergent validity.
Change in Advanced Clinical Solutions- Social Perception- Facial Affect Naming subscale (ACS-SP-FAN) | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (TBI participant only) In this affect recognition test, participants are shown 24 faces (different from ICARE training) that express happy, sad, angry, fearful, disgust, surprise or neutral emotions and must choose from a list of response options. The ACS-SP-FAN has good discriminant validity, high internal consistency, and high test-retest reliability.
Change in Brock Adaptive Functioning Questionnaire, empathy subscale (BAFQ-E) | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  This subjective measure, which has been designed for self and proxy ratings, includes several subscales (including empathy) to evaluate neurobehavioral functioning. Only the empathy subscale will be completed. Both the participant with TBI (self-rated) and their CP (about person with TBI). They will rate the frequency of occurrence of empathic behaviors on a 5-point scale. The BAFQ has high internal consistency, good concurrent validity with executive functioning measures, and correlates highly with caregiver stress and satisfaction, and return to work.
Change in Daily Empathic Behavior Survey (DEBS) | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (CP participant only) The DEBS was created for this study. For 1-week (7 days) intervals following each time frame point, CPs will be sent an electronic prompt to their cell phones at the end of the day and asked to rate the following statements on a scale from 1 (not at all) to 5 (extremely): Today, he/she 1) tried to understand others' thoughts, feelings, or problems; 2) considered others' perspectives and situations; 3) shared in others' feelings (e.g., felt sad with someone sad; felt happy with someone happy); 4) showed care and concern for others (e.g., asked, listened, comforted, consoled); 5) listened when others needed to talk; and 6) showed appreciation to others. If the CP did not interact with the participant that day, they will reply "no interaction" to that daily survey. While administered 7 times per time frame point/assessment period, the goal is a minimum of 3 completed surveys that period.
Change in Participation Assessment with Combined Tools-Objective (PART-O) | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (TBI participant only) PART-O is a standardized 17-item measure developed by the TBIMS to evaluate participation in the community with respect to three domains: Productivity, Social Relations, and Out and About. Items are scored on a 0 to 5 scale. Total PART-O scores will be used for our analyses.
Change in Global Impression of Change | Week 14, week 26, week 38
  Using a 7-point Likert scale, participants with TBI and CP will be asked to rate the degree of change (1=no change; 7=a great deal better) in a) overall functioning, b) empathy, and c) social behaviors of the person with TBI, as believed to be related to ICARE.
Change in Patient Reported Outcome Measurement Information System (PROMIS) Emotional Support Scale- modified | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (CP participant only) This 8-item subjective measure requires participants to rate the degree of emotional support they receive using a 5-point Likert scale. It will be completed by CP and modified to specifically inquire about the emotional support they receive from the participant with TBI (as opposed to support from anyone). PROMIS item banks and their short forms have been found to be reliable and precise measures that are comparable to legacy instruments.
Change in TBI CareQol Emotional Suppression- Short Form | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (CP participant only) Six items assess CP attempts to hide or suppress negative feelings in their caregiver role. Psychometric properties are strong.
Change in TBI CareQol Caregiver specific Anxiety | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  (CP participant only) This scale examines caregiver concerns about the person they care for with regard to behavior in public, mental health, mood, and fear for the future on a 5-point Likert-type scale ranging from 1 (Never) to 5 (Always). Scores are converted to a T-scale with a mean of 50 (SD=10). Higher scores indicate more anxiety. With rigorous development standards, it has been found to have strong psychometric properties.
Change in Unidimensional Relationship Closeness Scale | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  To be completed by participants with TBI and their CP, this 12-item self-report scale measures the closeness of social and personal relationships using a 7-point Likert scale from Strongly Disagree to Strongly Agree. Has good psychometric qualities.
Change in Relationship Quality Survey | Baseline (pre-test 1), week 7, week 14, week 26, week 38
  This brief survey uses a 10-point scale to rate the quality of their relationship (from very poor to outstanding). It will be completed both by the participant with the TBI and their CP.
Treatment Satisfaction | Week 14
  Participants with TBI and CP will complete a post-treatment survey regarding their satisfaction with content and with remote delivery of the therapy program, using a 9-point scale. For example, participants will be asked questions, such as: "Overall, how satisfied were you with ICARE therapy?" (Content satisfaction); and "How satisfied were you with receiving this type of treatment remotely/ via teletherapy?" (Teletherapy satisfaction). To guide future iterations, participants will be asked to describe 2-3 three things they liked, disliked and would change; and seek feedback on how the program could be improved.
Perth Empathy Scale (PES) | Week 7, week 14, week 26, week 38
  The Perth Empathy Scale (PES) is a subjective measure that evaluates general empathy ability that can be separated into cognitive and affective (negative and positive) empathy domains on a 5-point scale (1=Almost never; 5=Almost always). This subjective measure has also been designed to capture informant ratings, thus, both the participant with TBI (self-rated) and their CP (about person with TBI) will be assessed. Higher scores represent better empathic ability. Total scores range from 20-100; subscale scores range from 10-50 each. Participants will rate the frequency of occurrence in each behavior or experience. The PES has high convergent validity, discriminant validity in comparison to constructs like alexithymia, and criterion validity in assessing empathy in both positive and negative emotions.

CONTACTS AND LOCATIONS:
Overall Officials: Flora Hammond, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States